CLINICAL TRIAL: NCT04255927
Title: Triclosan-antibacterial Sutures Impact on the Incidence of Surgical Site Infection in Laparoscopic Sleeve Gastrectomy, Laparoscopic Appendectomy or Laparoscopic Cholecystectomy; Multi-center, Double-blind, Randomized Study.
Brief Title: Triclosan-antibacterial Sutures Impact on the Incidence of Surgical Site Infection in Laparoscopic Surgeries.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ClinAmygate (Other)
Collaborators: Misr University for Science and Technology (Other); Al Safwa Hospital (Unknown); Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Emad R Issak, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PR2019-26
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Laparoscopic Surgery; Surgical Wound; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection | interventions — Triclosan

STUDY DESIGN:
Intervention Model Description: randomized-controlled
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Coated Polyglactin 910 with Triclosan (Experimental): Coated Polyglactin 910 with Triclosan
  Interventions: Drug: Coated Vicryl plus
- Coated Polyglactin 910 without Triclosan (Active Comparator): Coated Polyglactin 910 without Triclosan
  Interventions: Drug: Coated vicryl

INTERVENTIONS:
Drug: Coated Vicryl plus — Vicryl plus (Coated Polyglactin 910 with Triclosan)
  Other Names: Coated Polyglactin 910 with Triclosan
  Arms: Coated Polyglactin 910 with Triclosan
Drug: Coated vicryl — Vicryl (Coated Polyglactin 910 without Triclosan)
  Other Names: Coated Polyglactin 910 without Triclosan
  Arms: Coated Polyglactin 910 without Triclosan

SUMMARY:
Comparing the incidence of PSI in cases using coated Polyglactin 910 suture with Triclosan and cases using Polyglactin 910 suture without Triclosan in laparoscopic sleeve gastrectomy, laparoscopic appendectomy or laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
In this prospective study, we will determine the incidence of PSI in Egypt as well as the impact of using coated polyglactin 910 sutures with Triclosan in lowering the incidence of PSI in laparoscopic sleeve gastrectomy, laparoscopic appendectomy or laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* candidate for laparoscopic surgical intervention during the period of the study were included.

Exclusion Criteria:

* Patient has immunodeficiency disorder.
* Patient receiving anti-cancer / immunosuppressive therapy.
* Patients with established pre-operative infection whether community acquired or hospital acquired either at / remote from the operative site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
port site infection (PSI) | 30 days
  the incidence of port site infection (PSI)

SECONDARY OUTCOMES:
hospital stay | 30 days
  Post-operative hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Emad R Issak, Diploma, Study Director — ClinAmygate
Locations (1):
- Misr Univeristy for Science and Technology Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmed I, Boulton AJ, Rizvi S, Carlos W, Dickenson E, Smith NA, Reed M. The use of triclosan-coated sutures to prevent surgical site infections: a systematic review and meta-analysis of the literature. BMJ Open. 2019 Sep 3;9(9):e029727. doi: 10.1136/bmjopen-2019-029727. PMID 31481559